CLINICAL TRIAL: NCT03212872
Title: Evaluation of Blood Ammonia Level as a Non Invasive Predictor for Presence of Gastroesophageal Varices and Risk of Bleeding
Brief Title: Blood Ammonia as Predictor for Esophageal Varices and Risk of Bleeding
Acronym: EV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ferial El-Kalla, Professor, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 30142/03/31
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Chronic Liver Disease; Esophageal Varices
Keywords: Ammonia; bleeding risk factors; endoscopic risk signs for bleeding; esophageal varices
MeSH Terms: conditions — Esophageal and Gastric Varices | interventions — Endoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopy (Other)
  Interventions: Diagnostic Test: Endoscopy

INTERVENTIONS:
Diagnostic Test: Endoscopy

SUMMARY:
Assessment of blood ammonia level as a non-invasive predictor for presence of EV and risk of bleeding

DETAILED DESCRIPTION:
A prospective cross sectional study on 150 consecutive patients screening for esophageal varices.

Patient groups groups:

Group (1): 100 patients with esophageal varices

Group (2): 50 chronic liver disease patients with no esophageal varices as a control group.

All patients will be subjected to:

1. - Detailed history-taking
2. - Full clinical examination
3. - Laboratory investigations:

   * Complete blood picture (CBC)
   * Erythrocyte sedimentation rate (ESR)
   * Renal function tests
   * Liver function tests
   * Prothrombin time and activity
   * Viral markers (HCV Ab - HBV Ag)
   * Blood ammonia level.
4. - Pelviabdominal US: Ultrasound examination of the liver, portal venous system, spleen, kidney and other abdominal organs.
5. - Upper GITendoscopy:

   * Varices will be classified according to the Japanese classification 1996,
   * The Baveno 11 score will be used to differentiate between mild and severe portal hypertensive gastropathy.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic liver disease

Exclusion Criteria:

* Patient in hepatic encephalopathy or coma.
* Patient in active bleeding or with history of bleeding within the two weeks prior to entry in the study .
* Patients with heart failure.
* Patients with renal failure.
* Patient with hepatocellular carcinoma and portal vein thrombosis.
* Patient taking Beta blockers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-07-07 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
level of serum ammonia in patients with risk factors for bleeding from esophageal varices | 24 months
  estimation of level of serum ammonia in patients with risk factors for bleeding from esophageal varices

CONTACTS AND LOCATIONS:
Overall Officials: Ferial El-Kalla, MD, Principal Investigator — Tanta University
Locations (1):
- Tanta Faculty of Medicine, Tanta, Gharbiah, Egypt